CLINICAL TRIAL: NCT02791373
Title: A Randomized Evaluation of Vinorelbine Versus Gemcitabine for Mobilization of Peripheral Stem Cells in Myeloma Patients Undergoing Autologous Stem Cell Transplantation.
Brief Title: Vinorelbine and Gemcitabine in Myeloma
Acronym: ViGeM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ViGeM
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Multiple Myeloma; Amyloidosis
MeSH Terms: conditions — Multiple Myeloma; Amyloidosis | interventions — Vinorelbine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobilisation Chemotherapy: Vinorelbine (Active Comparator): Vinorelbine is given at a standard dose of 35mg/m2 i.v. at day 1 as an infusion over 10 minutes, on an ambulatory basis.
  Interventions: Drug: Vinorelbine
- Mobilisation Chemotherapy: Gemcitabine (Experimental): Gemcitabine is given at the standard dose of 1250 mg/m2 i.v. in 500ml NaCl 0.9% (sodium chloride) as an infusion over 30 minutes, on an ambulatory basis.
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Vinorelbine — Mobilisation Chemotherapy
  Other Names: Navelbine
  Arms: Mobilisation Chemotherapy: Vinorelbine
Drug: Gemcitabine — Mobilisation Chemotherapy
  Other Names: Gemcitabine Sandoz
  Arms: Mobilisation Chemotherapy: Gemcitabine

SUMMARY:
The purpose of this study is to determine whether the efficacy of gemcitabine is comparable with the efficacy of the standard chemotherapy with vinorelbine for mobilization of autologous stem cells in myeloma patients

DETAILED DESCRIPTION:
Mobilization and engraftment of autologous peripheral blood progenitor cells (PBPC) in newly diagnosed multiple myeloma (MM) or amyloidosis patients followed by high dose chemotherapy with PBPC support.

Eligible are symptomatic myeloma or amyloidosis patients after standard first-line induction treatment. Patients must be fit for subsequent consolidation with high-dose chemotherapy with melphalan with autologous stem cell support.

Chemotherapy with vinorelbine is given at a standard dose of 35mg/m2 i.v. at day 1 as an infusion over 10 minutes, on an ambulatory basis. Gemcitabine is given at the standard dose of 1250 mg/m2 i.v. in 500ml NaCl 0.9% (sodium chlorid) as an infusion over 30 minutes, on an ambulatory basis.

G-CSF (granulocyte-colony stimulating factor) is given at 60 Mio s.c./d for patients ≤ 69kg in two daily doses of 30 Mio 12 hours apart, at 78 Mio s.c./d for patients from 70kg to 89kg with 48 Mio given in the morning and 30 Mio given in the evening, and at 96 Mio s.c./d for patients ≥ 90kg in two daily doses of 48 Mio.

Patients will be randomized in a 1:1 ratio between vinorelbine and gemcitabine mobilization. Patients will be stratified according to (A) response to induction treatment (refractory/stable disease/partial response versus very good partial response/complete response) and (B) peripheral neuropathy present versus absent before mobilization.

The high dose chemotherapy supported by autologous stem cell transplantation is not part of the study treatment. Standard high dose melphalan (200 mg/m2) will be used as conditioning regimen. After transplantation, G-CSF will be given to subjects starting at day +6 until day +11 after PBPC re-infusion, at a dose of 30 Mio per day for patients ≤ 75kg, and of 48 Mio for patients >75kg.

Planned accrual is chemotherapy with vinorelbine is given at a standard dose of 35mg/m2 i.v. at day 1 as an infusion over 10 minutes, on an ambulatory basis. Gemcitabine is given at the standard dose of 1250 mg/m2 i.v. in 500ml NaCl 0.9% as an infusion over 30 minutes, on an ambulatory basis.

G-CSF is given at 60 Mio s.c./d for patients ≤ 69kg in two daily doses of 30 Mio 12 hours apart, at 78 Mio s.c./d for patients from 70kg to 89kg with 48 Mio given in the morning and 30 Mio given in the evening, and at 96 Mio s.c./d for patients ≥ 90kg in two daily doses of 48 Mio.

Patients will be randomized in a 1:1 ratio between vinorelbine and gemcitabine mobilization. Patients will be stratified according to (A) response to induction treatment (refractory/stable disease/partial response versus very good partial response/complete response) and (B) peripheral neuropathy present versus absent before mobilization.

The high dose chemotherapy supported by autologous stem cell transplantation is not part of the study treatment. Standard high dose melphalan (200 mg/m2) will be used as conditioning regimen. After transplantation, G-CSF will be given to subjects starting at day +6 until day +11 after PBPC re-infusion, at a dose of 30 Mio per day for patients ≤ 75kg, and of 48 Mio for patients >75kg.

Planed accrual of 136 patients in 42 months.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic myeloma or amyloidosis patients after standard first-line induction treatment. Patients must be fit for subsequent consolidation with high-dose chemotherapy with melphalan with autologous stem cell support.
* Standard induction chemotherapy comprises regimens including thalidomide, bortezomib, or lenalidomide (less than 5 cycles), alone or in combination with dexamethasone. Combinations of novel agents are allowed as well as induction with the VAD (vincristine, adriamycin and dexamethasone) regimen.
* Patient must be aged 18-75 years, with an ECOG (Eastern Cooperative Oncology Group) < 3, and has given voluntary written informed consent.
* Patient has the following laboratory values at baseline:
* Platelets count > 50 x 109/l without transfusion support within 7 days before the laboratory test.
* Absolute neutrophil count (ANC) > 1.0 x 109/l without the use of colony stimulating factors.
* Creatinine-clearance > 40 ml/min
* Negative pregnancy test (urine or serum) within 14 days prior to registration for all women of childbearing potential. Patients of childbearing potential must implement adequate measures (hormonal treatment p.o. or i.m., intra uterine surgical devices, or latex condoms) to avoid pregnancy during study treatment and for additional 12 months. No pregnant or lactating patients are allowed.

Exclusion Criteria:

* Patients with more than 4 cycles of chemotherapy with lenalidomide.
* Patients not fit for autologous stem cell transplantation
* Patients with other serious medical condition that could potentially interfere with the completion of treatment according to this protocol or that would impair tolerance to therapy or prolong hematological recovery.
* Subject is currently enrolled in another investigational trial or is receiving other investigational agent(s).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2014-03; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
CD34+ (cluster of differentiation 34) peripheral blood stem cells | Day 8
  Number of patients with collection of > 6 million CD34+ peripheral blood stem cells/kg body weight at day 8 after vinorelbine versus gemcitabine chemotherapy

SECONDARY OUTCOMES:
Rate of peripheral neuropathy | Between 15 and 30 days
  Number of patients with peripheral neuropathy following mobilization chemotherapy with vinorelbine versus gemcitabine. Clinical assessment will be done between 15 and 30 days after autologous transplant
Severity of peripheral neuropathy | Between 15 and 30 days
  Grade of peripheral neuropathy following mobilization chemotherapy with vinorelbine versus gemcitabine. Clinical assessment will be done between 15 and 30 days after autologous transplant
Hematologic recovery | Between 15 and 30 days
  Time (days) until hematologic recovery (Leucocytes > 3.0 G/L and Thrombocytes >100 G/L) following autologous transplantation comparing patients mobilized with vinorelbine versus gemcitabine.
Minimal residual disease in the peripheral blood | Day 8
  Minimal residual disease in the peripheral blood at the day of stem cell collection (day 8) using flow cytometry multiparameter assessment comparing patients mobilized with vinorelbine versus gemcitabine.
Need to use the stem cell releasing compound Plerixafor | Day 8
  Number of patients who needs to use the stem cell releasing compound Plerixafor at day 9 in patients with insufficient peripheral stem cell mobilization (at day 8) comparing patients mobilized with vinorelbine versus gemcitabine.
Response Rate | Between 15 and 30 days
  Response (myeloma parameter) to the mobilization chemotherapy comparing patients mobilized with vinorelbine versus gemcitabine.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pabst, MD, Study Chair — Inselspital , University Hospital Berne
Locations (1):
- Department for Medical Oncology; University Hospital/Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Attal M, Harousseau JL, Stoppa AM, Sotto JJ, Fuzibet JG, Rossi JF, Casassus P, Maisonneuve H, Facon T, Ifrah N, Payen C, Bataille R. A prospective, randomized trial of autologous bone marrow transplantation and chemotherapy in multiple myeloma. Intergroupe Francais du Myelome. N Engl J Med. 1996 Jul 11;335(2):91-7. doi: 10.1056/NEJM199607113350204. PMID 8649495